CLINICAL TRIAL: NCT03976323
Title: A Phase 3 Study of Pembrolizumab in Combination With Pemetrexed/Platinum (Carboplatin or Cisplatin) Followed by Pembrolizumab and Maintenance Olaparib vs Maintenance Pemetrexed in the First-Line Treatment of Participants With Metastatic Nonsquamous Non-Small-Cell Lung Cancer (NSCLC)
Brief Title: Study of Pembrolizumab With Maintenance Olaparib or Maintenance Pemetrexed in First-line (1L) Metastatic Nonsquamous Non-Small-Cell Lung Cancer (NSCLC) (MK-7339-006, KEYLYNK-006)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7339-006; MK-7339-006 (Other: MSD); KEYLYNK-006 (Other: MSD); 194895 (Registry Identifier: JAPIC-CTI); 2023-509774-40-00 (Registry Identifier: EU CT); U1111-1300-7107 (Registry Identifier: UTN); 2018-004720-11 (EudraCT Number)
Record Dates: First submitted 2019-06-03; First posted 2019-06-06 (Actual); Results first posted 2025-02-06 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Carcinoma, Nonsquamous Non-small-cell Lung
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Cell Death 1 Ligand 1 (PDL1, PD-L1); Programmed Cell Death 1 Ligand 2 (PDL2, PD-L2)
MeSH Terms: conditions — Carcinoma; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Pemetrexed; Carboplatin; Cisplatin; olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab + Pemetrexed + Platinum Therapy + Olaparib (Experimental): For the Induction Phase, participants receive 4 cycles (up to ~12 weeks [cycle = 3 weeks]): pembrolizumab 200 mg intravenous (IV) on Day 1 of each cycle (cycles 1 through 4) PLUS pemetrexed 500 mg/m^2 IV on Day 1 of each cycle (cycles 1 through 4) PLUS platinum chemotherapy, investigator's choice: carboplatin area under the curve (AUC) 5 mg/mL/min IV on Day 1 of each cycle (Cycles 1 through 4) OR cisplatin 75 mg/m^2 IV on Day 1 of each cycle (Cycles 1 through 4).
  If the participant has a complete/partial response or stable disease to induction therapy, the participant can enter the Maintenance Phase and receive pembrolizumab 200 mg IV on Day 1 of each 3-week cycle for up to 31 cycles PLUS maintenance oral olaparib 300 mg twice daily. The participant can continue to receive maintenance olaparib until progressive disease or toxicity. Across both phases, participants can receive pembrolizumab for a total treatment duration of up to ~35 cycles (up to ~2 years [cycle = 3 weeks]).
  Interventions: Biological: Pembrolizumab; Drug: Pemetrexed; Drug: Carboplatin; Drug: Cisplatin; Drug: Olaparib
- Pembrolizumab + Pemetrexed + Platinum Therapy + Pemetrexed (Active Comparator): For the Induction Phase, participants receive 4 cycles (up to ~12 weeks [cycle = 3 weeks]): pembrolizumab 200 mg IV on Day 1 of each cycle (cycles 1 through 4) PLUS pemetrexed 500 mg/m^2 IV on Day 1 of each cycle (cycles 1 through 4) PLUS platinum chemotherapy, investigator's choice: carboplatin AUC 5 mg/mL/min IV on Day 1 of each cycle (Cycles 1 through 4) OR cisplatin 75 mg/m^2 IV on Day 1 of each cycle (Cycles 1 through 4).
  If the participant has a complete/partial response or stable disease to induction therapy, the participant can enter the Maintenance Phase and receive pembrolizumab 200 mg IV on Day 1 of each 3-week cycle for up to 31 cycles PLUS maintenance pemetrexed 500 mg/m^2 IV on Day 1 of each 3-week cycle. The participant can continue to receive maintenance pemetrexed until progressive disease or toxicity. Across both phases, participants can receive pembrolizumab for a total treatment duration of up to ~35 cycles (up to ~2 years [cycle = 3 weeks]).
  Interventions: Biological: Pembrolizumab; Drug: Pemetrexed; Drug: Carboplatin; Drug: Cisplatin

INTERVENTIONS:
Biological: Pembrolizumab — IV infusion
  Other Names: MK-3475; KEYTRUDA®
Drug: Pemetrexed — IV infusion
  Other Names: ALIMTA®
Drug: Carboplatin — IV infusion
  Other Names: PARAPLATIN®
Drug: Cisplatin — IV infusion
  Other Names: PLATINOL®; PLATINOL®-AQ
Drug: Olaparib — Oral Tablet
  Other Names: LYNPARZA®
  Arms: Pembrolizumab + Pemetrexed + Platinum Therapy + Olaparib

SUMMARY:
The current study will compare pembrolizumab (MK-3475) plus maintenance olaparib, versus (vs) pembrolizumab plus maintenance pemetrexed for the treatment of non-squamous NSCLC. The study's 2 primary hypotheses are: 1. Pembrolizumab plus maintenance olaparib is superior to pembrolizumab plus maintenance pemetrexed with respect to progression-free survival (PFS) per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) by blinded independent clinical review (BICR) and 2. Pembrolizumab plus maintenance olaparib is superior to pembrolizumab plus maintenance pemetrexed with respect to overall survival (OS).

DETAILED DESCRIPTION:
This study has 2 phases: an Induction Phase of up to ~4 Cycles (up to ~12 weeks [cycle =3 weeks]) and a Maintenance Phase of up to ~31 cycles of pembrolizumab (cycle = 3 weeks]); total pembrolizumab treatment duration will be up to ~35 cycles (up to ~2 years). In the Induction Phase, participants receive pembrolizumab plus pemetrexed plus platinum (carboplatin or cisplatin, at the investigator's discretion). In the Maintenance Phase, participants with a partial or complete disease response or with stable disease after completing four cycles of induction therapy and who meet eligibility criteria will be randomly assigned to receive pembrolizumab plus maintenance olaparib OR pembrolizumab plus maintenance pemetrexed. In the Maintenance Phase, participants receive pembrolizumab for up to 31 cycles (cycle = 3 weeks) plus maintenance olaparib OR maintenance pemetrexed until progressive disease (PD), intolerable toxicities, or physician decision.

Qualified participants in each study arm of the maintenance phase (Pembrolizumab plus Olaparib and Pembrolizumab plus Pemetrexed) who complete up to ~35 cycles of pembrolizumab (up to ~2 years [cycle =3 weeks]) may be eligible to receive a second course of pembrolizumab for up to ~17 cycles (up to ~1 additional year). Per protocol, response or progression during the second pembrolizumab course will not be counted towards patient reported outcomes (PROs) or efficacy outcome measures and adverse events during the second pembrolizumab course will not be counted towards safety outcome measures.

ELIGIBILITY:
Inclusion Criteria:

1. Have a histologically or cytologically confirmed diagnosis nonsquamous NSCLC.
2. Have stage IV nonsquamous NSCLC.
3. Have confirmation that epidermal growth factor receptor (EGFR), anaplastic lymphoma kinase (ALK), or Proto-oncogene tyrosine-protein kinase (ROS1)-directed therapy is not indicated.
4. Have measurable disease based on RECIST 1.1.
5. Have provided archival tumor tissue sample or newly obtained core or incisional biopsy of a tumor lesion not previously irradiated.

   Note: Adequacy of biopsy specimen for the above analyses must be confirmed by the central laboratory before the participant can start the induction phase. Submission of another tumor specimen may be required prior to enrolling the participant, if adequate tumor tissue was not provided the first time.
6. Have a life expectancy of at least 3 months.
7. Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Status assessed within 7 days prior to the administration of study intervention.
8. Have not received prior systemic treatment for their advanced/metastatic NSCLC.
9. Have adequate organ function.
10. Male and female participants who are not pregnant and of childbearing potential must follow contraceptive guidance during the treatment period and for 180 days afterwards.
11. Male participants must refrain from donating sperm, and female participants must refrain from donating eggs to others or freeze/store for her own use during the treatment period and for 180 days afterwards.

Exclusion Criteria:

1. Has predominantly squamous cell histology NSCLC.
2. Has a known additional malignancy that is progressing or has progressed within the past 3 years requiring active treatment.
3. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
4. Has a severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
5. Has a known hypersensitivity to any components or excipients of cisplatin, carboplatin, pemetrexed, or olaparib.
6. Has an active autoimmune disease that has required systemic treatment in past 2 years.
7. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy.
8. Has a known history of human immunodeficiency virus (HIV) infection, a known history of hepatitis B infection, or known active hepatitis C virus infection.
9. Has interstitial lung disease, or history of pneumonitis requiring systemic steroids for treatment.
10. Has received prior therapy with olaparib or with any other polyadenosine 5' diphosphoribose (polyADP ribose) polymerization (PARP) inhibitor.
11. Has received prior therapy with an agent directed to programmed cell death ligand 1 (PD-L1), anti PD-L2, or directed to a stimulatory or co-inhibitory T-cell receptor (e.g., cytotoxic T-lymphocyte-associated protein 4 (CTLA-4), OX-40, CD137).
12. Has myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML) or with features suggestive of MDS/AML.
13. Has history of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 2 years.
14. Has completed palliative radiotherapy within 7 days of the first dose. Participants must have recovered from all radiation-related toxicities and not require corticosteroids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1003 (Actual)
Dates: Start 2019-06-28 (Actual); Primary Completion 2024-02-07 (Actual); Study Completion 2026-01-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (178):
- United States (20):
  - Alabama Oncology Bruno Cancer Center ( Site 0001), Birmingham, Alabama
  - Northwest Alabama Cancer Center, PC ( Site 0002), Muscle Shoals, Alabama
  - Disney Family Cancer Center ( Site 0005), Burbank, California
  - Boca Raton Regional Hospital ( Site 0018), Boca Raton, Florida
  - Mid-Florida Cancer Centers ( Site 0022), Orange City, Florida
  - Moffitt Cancer Center ( Site 0024), Tampa, Florida
  - Columbus Regional Research Institute ( Site 0098), Columbus, Georgia
  - Mount Sinai Hospital Medical Center ( Site 0032), Chicago, Illinois
  - Oncology of Northshore ( Site 0033), Rolling Meadows, Illinois
  - Methodists Hospitals/Premier Oncology Hematology Associates ( Site 0036), Merrillville, Indiana
  - Medstar Good Samaritan Hospital ( Site 0040), Baltimore, Maryland
  - Barbara Ann Karmanos Cancer Institute ( Site 0041), Detroit, Michigan
  - Hattiesburg Clinic ( Site 0045), Hattiesburg, Mississippi
  - Frontier Oncology ( Site 0080), Billings, Montana
  - Bozeman Health Deaconness Cancer Center ( Site 0046), Bozeman, Montana
  - Waverly Hematology Oncology ( Site 0081), Cary, North Carolina
  - Thompson Cancer Survival Center ( Site 2812), Knoxville, Tennessee
  - University of Tennessee Medical Center Knoxville ( Site 0060), Knoxville, Tennessee
  - Renovatio Clinical ( Site 0062), The Woodlands, Texas
  - Cancer Care Northwest ( Site 0071), Spokane Valley, Washington
- Argentina (8):
  - Hospital Italiano Regional del Sur ( Site 0509), Bahía Blanca, Buenos Aires
  - Hospital Italiano de Buenos Aires-Clinical Oncology ( Site 0511), Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Hospital Britanico de Buenos Aires ( Site 0500), Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Instituto Medico Rio Cuarto ( Site 0501), Río Cuarto, Córdoba Province
  - Centro Oncológico de Rosario ( Site 0507), Rosario, Santa Fe Province
  - Centro Medico San Roque ( Site 0506), San Miguel de Tucumán, Tucumán Province
  - Clínica Universitaria Reina Fabiola ( Site 0505), Córdoba
  - Sanatorio Privado San Geronimo S.R.L ( Site 0510), Santa Fe
- Australia (4):
  - Liverpool Hospital ( Site 1201), Liverpool, New South Wales
  - Southern Medical Day Care Centre ( Site 1200), Wollongong, New South Wales
  - Townsville General Hospital ( Site 1202), Townsville, Queensland
  - Monash Cancer Centre ( Site 1205), Clayton, Victoria
- Austria (5):
  - Innsbruck LKH ( Site 1302), Innsbruck, Tyrol
  - Ordensklinikum Linz GmbH Elisabethinen ( Site 1307), Linz, Upper Austria
  - Klinikum Wels-Grieskirchen ( Site 1304), Wels, Upper Austria
  - Social Medical Center - Otto Wagner Hospital ( Site 1301), Vienna, Vienna
  - Krankenhaus Nord - Klinik Floridsdorf ( Site 1300), Vienna
- Brazil (14):
  - Instituto do Cancer do Ceara ( Site 0201), Fortaleza, Ceará
  - Hospital Sao Rafael ( Site 0212), Salvador, Estado de Bahia
  - Oncologica do Brasil ( Site 0210), Belém, Pará
  - Hospital Tacchini ( Site 0208), Bento Gonçalves, Rio Grande do Sul
  - Irmandade da Santa Casa de Misericordia de Porto Alegre ( Site 0209), Porto Alegre, Rio Grande do Sul
  - Saint Gallen Instituto de Oncologia ( Site 0206), Santa Cruz do Sul, Rio Grande do Sul
  - YNOVA Pesquisa Clinica ( Site 0215), Florianópolis, Santa Catarina
  - Centro de Novos Tratamentos Itajai - Clinica de Neoplasias Litoral ( Site 0202), Itajaí, Santa Catarina
  - Centro de Hematologia e Oncologia ( Site 0205), Joinville, Santa Catarina
  - Hospital de Base de Sao Jose de Rio Preto ( Site 0204), Sao Jose Rio Preto, São Paulo
  - Instituto Nacional do Cancer Jose Alencar Gomes da Silva INCA ( Site 0203), Rio de Janeiro
  - Instituto do Cancer do Estado de Sao Paulo - ICESP ( Site 0200), São Paulo
  - BP - A Beneficencia Portuguesa de São Paulo-Medical Oncology ( Site 0214), São Paulo
  - Hospital Paulistano - Amil Clinical Research ( Site 0207), São Paulo
- Canada (11):
  - Lions Gate Hospital ( Site 0106), North Vancouver, British Columbia
  - BC Cancer - Victoria ( Site 0109), Victoria, British Columbia
  - Queen Elizabeth II Health Sciences Centre ( Site 0107), Halifax, Nova Scotia
  - Health Sciences North Research Institute ( Site 0115), Greater Sudbury, Ontario
  - Waterloo Regional Health Network (WRHN) ( Site 0117), Kitchener, Ontario
  - Stronach Regional Cancer Centre ( Site 0101), Newmarket, Ontario
  - CISSS de la Monteregie-Centre ( Site 0114), Greenfield Park, Quebec
  - Centre Hospitalier de l Universite de Montreal - CHUM ( Site 0105), Montreal, Quebec
  - CIUSSS Ouest de l Ile - St-Mary s Hospital ( Site 0110), Montreal, Quebec
  - Centre de Sante et des Services Sociaux de Rimouski-Neigette ( Site 0104), Rimouski, Quebec
  - CIUSSS de l Estrie - CHUS - Centre Hosp. Univ. Sherbrooke ( Site 0103), Sherbrooke, Quebec
- Colombia (4):
  - Fundacion Colombiana de Cancerologia Clinica Vida ( Site 0604), Medellín, Antioquia
  - Clinica de la Costa S.A.S. ( Site 0608), Barranquilla, Atlántico
  - Administradora Country S.A. ( Site 0603), Bogotá, Bogota D.C.
  - Clinica Colsanitas S.A. Sede Clinica Universitaria Colombia ( Site 0601), Bogotá, Bogota D.C.
- France (9):
  - Institut De Cancerologie De Lorraine ( Site 1409), Vandœuvre-lès-Nancy, Ain
  - Centre Hospitalier De Chauny ( Site 1411), Chauny, Aisne
  - CHU Caen ( Site 1406), Caen, Calvados
  - CHU Angers ( Site 1405), Angers, Maine-et-Loire
  - Hopital Robert Schuman ( Site 1402), Vantoux, Moselle
  - Centre Jean Perrin ( Site 1407), Clermont-Ferrand, Puy-de-Dome
  - Centre Hospitalier de Pau ( Site 1412), Pau, Pyrenees-Atlantiques
  - CHU de Rouen ( Site 1403), Rouen, Seine-Maritime
  - Hopital d'Instruction des Armees Begin ( Site 1413), Saint-Mandé, Val-de-Marne
- Germany (13):
  - Studienzentrum Aschaffenburg ( Site 1525), Aschaffenburg, Bavaria
  - Klinikum der LMU ( Site 1500), Munich, Bavaria
  - Klinikum Bogenhausen Staedt. Klinikum Muenchen GmbH ( Site 1523), Munich, Bavaria
  - Universitaetsklinikum Regensburg ( Site 1512), Regensburg, Bavaria
  - Klinikum Wuerzburg Mitte gGmbH ( Site 1509), Würzburg, Bavaria
  - Universitaetsklinikum Frankfurt ( Site 1513), Frankfurt am Main, Hesse
  - Pneumologische Lehrklinik Universitaet Goettingen ( Site 1501), Immenhausen, Hesse
  - Universitaetsmedizin Goettingen ( Site 1507), Göttingen, Lower Saxony
  - Universitaetsklinikum Bonn ( Site 1524), Bonn, North Rhine-Westphalia
  - Kliniken Essen Mitte ( Site 1517), Essen, North Rhine-Westphalia
  - InVo-Institut fuer Versorgungsforschung in der Onkologie ( Site 1514), Koblenz, Rhineland-Palatinate
  - Helios Klinikum Erfurt GmbH ( Site 1502), Erfurt, Thuringia
  - Katholisches Marienkrankenhaus gGmbH ( Site 1522), Hamburg
- Japan (14):
  - National Hospital Organization Nagoya Medical Center ( Site 0806), Nagoya, Aichi-ken
  - Aichi Cancer Center ( Site 0803), Nagoya, Aichi-ken
  - National Cancer Center Hospital East ( Site 0801), Kashiwa, Chiba
  - Kanazawa University Hospital ( Site 0811), Kanazawa, Ishikawa-ken
  - Kanagawa Cancer Center ( Site 0807), Yokohama, Kanagawa
  - Sendai Kousei Hospital ( Site 0812), Sendai, Miyagi
  - Kansai Medical University Hospital ( Site 0804), Hirakata, Osaka
  - National Hospital Organization Kinki-chuo Chest Medical Center ( Site 0813), Sakai, Osaka
  - Shizuoka Cancer Center ( Site 0802), Suntogun, Shizuoka
  - National Hospital Organization Kyushu Medical Center ( Site 0805), Fukuoka
  - Niigata Cancer Center Hospital ( Site 0808), Niigata
  - Okayama University Hospital ( Site 0810), Okayama
  - Osaka International Cancer Institute ( Site 0809), Osaka
  - Cancer Institute Hospital of JFCR ( Site 0800), Tokyo
- New Zealand (2):
  - MidCentral DHB Palmerston North Hospital ( Site 1102), Palmerston North, Manawatu-Wanganui
  - Capital & Coast District Health Board - Wellington Hospital ( Site 1101), Wellington
- Poland (7):
  - Przychodnia Lekarska Komed ( Site 2416), Konin, Greater Poland Voivodeship
  - MED-POLONIA Sp. z o.o. ( Site 2419), Poznan, Greater Poland Voivodeship
  - Krakowski Szpital Specjalistyczny im Jana Pawla II ( Site 2420), Krakow, Lesser Poland Voivodeship
  - Wielospecjalistyczny Szpital SPZOZ w Zgorzelcu ( Site 2404), Zgorzelec, Lower Silesian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy w Warszawie ( Site 2418), Warsaw, Masovian Voivodeship
  - Szpital Rejonowy im. dr Jozefa Rostka ( Site 2402), Racibórz, Silesian Voivodeship
  - Warminsko-Mazurskie Centrum Chorob Pluc w Olsztynie ( Site 2417), Olsztyn, Warmian-Masurian Voivodeship
- Romania (7):
  - MEMORIAL HEALTHCARE INTERNATIONAL S.R.L. ( Site 2502), Bucharest, București
  - Cardiomed SRL Cluj-Napoca ( Site 2504), Cluj-Napoca, Cluj
  - S.C. Radiotherapy Center Cluj S.R.L ( Site 2507), Cluj-Napoca, Cluj
  - Ovidius Clinical Hospital OCH ( Site 2501), Ovidiu, Constanța County
  - S.C. Centrul de Oncologie Sf. Nectarie SRL ( Site 2508), Craiova, Dolj
  - Policlinica Oncomed SRL ( Site 2505), Timișoara, Timiș County
  - Spitalul PDR Medlife ( Site 2509), Brasov
- Russia (13):
  - Russian Oncological Research Center n.a. N.N.Blokhin of MoH ( Site 2000), Moscow, Moscow
  - First Moscow State Medical University n.a. I.M.Sechenov ( Site 2024), Moscow, Moscow
  - Moscow Research Oncology Institute named after P.A. Hertsen ( Site 2009), Moscow, Moscow
  - FSAI Treatment and Rehabilitation Centre of the MoH and SD of RF ( Site 2006), Moscow, Moscow
  - Moscow Regional Oncological Dispensary ( Site 2028), Balashikha, Moscow Oblast
  - Nizhniy Novgorod Region Oncology Dispensary ( Site 2026), Nizhny Novgorod, Nizhny Novgorod Oblast
  - Budgetary Healthcare Institution of Omsk Region Clinical Oncology Dispensary-Chemotherapy #1 ( Site 2010), Omsk, Omsk Oblast
  - SBHI Samara Regional Clinical Oncology Dispensary ( Site 2016), Samara, Samara Oblast
  - SBHI Leningrad Regional Clinical Hospital ( Site 2002), Saint Petersburg, Sankt-Peterburg
  - SPb Central Clinical Railway Hospital ( Site 2003), Saint Petersburg, Sankt-Peterburg
  - National Medical Research Center of Oncology N.A. N.N. Petrov ( Site 2004), Saint Petersburg, Sankt-Peterburg
  - SPb SBHI City Clinical Oncological Dispensary ( Site 2001), Saint Petersburg, Sankt-Peterburg
  - Republican Clinical Oncology Dispensary of Tatarstan MoH named after professor M.Z. Sigal ( Site 2021), Kazan', Tatarstan, Respublika
- South Korea (8):
  - National Cancer Center ( Site 1006), Goyang-si, Kyonggi-do
  - The Catholic University of Korea St. Vincent s Hospital ( Site 1003), Suwon, Kyonggi-do
  - Ajou University Hospital ( Site 1004), Suwon, Kyonggi-do
  - Gyeongsang National University Hospital ( Site 1005), Jinju, Kyongsangnam-do
  - Chungbuk National University Hospital ( Site 1002), Cheongju-si, North Chungcheong
  - Asan Medical Center ( Site 1007), Songpa-gu, Seoul
  - Seoul National University Hospital ( Site 1000), Seoul
  - Korea University Guro Hospital ( Site 1008), Seoul
- Spain (5):
  - Hospital Universitario Quiron Madrid ( Site 1701), Pozuelo de Alarcón, Madrid
  - Hospital Clinico Universitario de Valencia ( Site 1706), Valencia, Valenciana, Comunitat
  - Hospital del Mar ( Site 1702), Barcelona
  - Hospital Universitario Nuestra Senora de Valme ( Site 1703), Seville
  - Hospital Clinico Lozano Blesa ( Site 1700), Zaragoza
- Taiwan (6):
  - Chang Gung Medical Foundation. Kaohsiung Branch ( Site 0907), Kaohsiung City
  - China Medical University Hospital ( Site 0904), Taichung
  - National Cheng Kung University Hospital ( Site 0905), Tainan
  - National Taiwan University Hospital ( Site 0900), Taipei
  - Mackay Memorial Hospital ( Site 0902), Taipei
  - Chang Gung Medical Foundation.Linkou Branch ( Site 0903), Taoyuan District
- Turkey (Türkiye) (9):
  - Namik Kemal Universitesi Tip Fakultesi ( Site 2100), Tekirdağ, Tekirdas
  - Baskent Unv. Adana Uyg. ve Arast. Hastanesi ( Site 2101), Adana
  - Gazi Universitesi Tip Fakultesi ( Site 2104), Ankara
  - Ankara Bilkent Sehir Hastanesi ( Site 2105), Ankara
  - Bezmialem Vakif Univ. Tıp Fakultesi Hastanesi Tibbi Onkoloji Bolumu ( Site 2107), Istanbul
  - Göztepe Prof. Dr. Süleyman Yalçın Şehir Hastanesi-oncology ( Site 2103), Istanbul
  - Ege Universitesi Tip Fakultesi ( Site 2109), Izmir
  - Erciyes Universitesi Tip Fakultesi ( Site 2108), Kayseri
  - Ondokuz Mayıs Universitesi-Oncology department ( Site 2106), Samsun
- Ukraine (12):
  - Cherkasy Regional Oncology Dispensary ( Site 2211), Cherkasy, Cherkasy Oblast
  - Municipal Non-Profit Enterprise City Clinical Hospital 4 of Dnipro City Council ( Site 2201), Dnipro, Dnipropetrovsk Oblast
  - MI Precarpathian Clinical Oncology Center ( Site 2204), Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - Grigoriev Institute for medical Radiology NAMS of Ukraine ( Site 2212), Kharkiv, Kharkivs’ka Oblast’
  - CNPE "Regional Center of Oncology"-Thoracic organs ( Site 2205), Kharkiv, Kharkivs’ka Oblast’
  - PP PPC Acinus Medical and Diagnostic Centre ( Site 2209), Kropyvnitskiy, Kirovohrad Oblast
  - Medical Center Asklepion LLC ( Site 2234), Khodosovka, Kyivska Oblast
  - Medical Center Verum ( Site 2230), Kyiv, Kyivska Oblast
  - Medical and Diagnostic Centre LLC Dobryi Prognoz ( Site 2213), Kyiv, Kyivska Oblast
  - MI Odessa Regional Oncological Centre ( Site 2208), Odesa, Odesa Oblast
  - Central City Clinical Hospital ( Site 2207), Uzhhorod, Zakarpattia Oblast
  - Kyiv City Clinical Oncology Centre ( Site 2210), Kyiv
- United Kingdom (7):
  - Barts Health NHS Trust - St Bartholomew s Hospital ( Site 1923), London, London, City of
  - Chelsea and Westminster Hospital ( Site 1901), London, London, City of
  - West Suffolk Hospitals NHS Trust ( Site 1919), Bury St Edmunds, Suffolk
  - Western General Hospital, Edinburgh ( Site 1924), Edinburgh, United Kingdom
  - Singleton Hospital ( Site 1909), Swansea, Wales
  - Colchester General Hospital ( Site 1911), Colchester, Worcestershire
  - Birmingham Heartlands Hospital ( Site 1910), Birmingham

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Result] Gray JE, Schenker M, Sendur MAN, Leonova V, Kowalski D, Kato T, Orlova R, Yang JC, Langleben A, Pilz A, Ungureanu A, Mak MP, De Angelis F, Aggarwal H, Zimmer Z, Zhao B, Shamoun M, Kim TM. The Phase 3 KEYLYNK-006 Study of Pembrolizumab Plus Olaparib Versus Pembrolizumab Plus Pemetrexed as Maintenance Therapy for Metastatic Nonsquamous NSCLC. J Thorac Oncol. 2025 Feb;20(2):219-232. doi: 10.1016/j.jtho.2024.10.026. Epub 2024 Nov 7. PMID 39521434
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26268&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Per protocol, response or progression during the second pembrolizumab course were not counted towards patient reported outcomes (PROs) or efficacy outcome measures and adverse events during the second pembrolizumab course will not be counted towards safety outcome measures.
Groups:
- Pembrolizumab + Pemetrexed + Platinum Therapy (Induction Phase): Participants received 4 cycles (up to ~12 weeks [cycle = 3 weeks]): pembrolizumab 200 mg intravenous (IV) on Day 1 of each cycle (cycles 1 through 4) PLUS pemetrexed 500 mg/m^2 IV on Day 1 of each cycle (cycles 1 through 4) PLUS platinum chemotherapy, investigator's choice: carboplatin area under the curve (AUC) 5 mg/mL/min IV on Day 1 of each cycle (Cycles 1 through 4) OR cisplatin 75 mg/m^2 IV on Day 1 of each cycle (Cycles 1 through 4).
- Pembrolizumab + Olaparib (Maintenance Phase): Eligible participants with a complete/partial response or stable disease to treatment in the Induction Phase could enter Maintenance Phase. For the Maintenance Phase, participants received pembrolizumab 200 mg IV on Day 1 of each 3-week cycle for up to 31 cycles PLUS maintenance oral olaparib 300 mg twice daily. In the Maintenance Phase, participants continued to receive maintenance olaparib until progressive disease or toxicity. Across both phases, participants could receive pembrolizumab for a total treatment duration of up to ~35 cycles (up to ~2 years [cycle = 3 weeks]). Qualified participants who completed up to ~35 cycles of pembrolizumab (up to ~2 years) may have been eligible to receive a second course of pembrolizumab at the same dose and schedule (200 mg on Day 1 of each 3-week cycle) for up to ~17 cycles (up to ~1 additional year).
- Pembrolizumab + Pemetrexed (Maintenance Phase): Eligible participants with a complete/partial response or stable disease to treatment in the Induction Phase could enter the Maintenance Phase. For the Maintenance Phase, participants received pembrolizumab 200 mg IV on Day 1 of each 3-week cycle for up to 31 cycles PLUS maintenance pemetrexed 500 mg/m^2 IV on Day 1 of each 3-week cycle. In the Maintenance Phase, participants continued to receive maintenance pemetrexed until progressive disease or toxicity. Across both phases, participants could receive pembrolizumab for a total treatment duration of up to ~35 cycles (up to ~2 years [cycle = 3 weeks]). Qualified participants who completed up to ~35 cycles of pembrolizumab (up to ~2 years) may have been eligible to receive a second course of pembrolizumab at the same dose and schedule (200 mg on Day 1 of each 3-week cycle) for up to ~17 cycles (up to ~1 additional year).
Period: Induction Phase
Arm/Group | Pembrolizumab + Pemetrexed + Platinum Therapy (Induction Phase) | Pembrolizumab + Olaparib (Maintenance Phase) | Pembrolizumab + Pemetrexed (Maintenance Phase)
Started | 1003 | 0 | 0
Completed | 672 | 0 | 0
Not Completed | 331 | 0 | 0
Not completed — Failure to Meet Maintenance Randomization Criteria | 251 | 0 | 0
Not completed — Death | 80 | 0 | 0
Period: Maintenance Phase
Arm/Group | Pembrolizumab + Pemetrexed + Platinum Therapy (Induction Phase) | Pembrolizumab + Olaparib (Maintenance Phase) | Pembrolizumab + Pemetrexed (Maintenance Phase)
Started | 0 | 337 (Per protocol, eligible participants were randomized to one of the maintenance treatment arms. Not all participants from the induction period continued into the randomized maintenance phase.) | 335 (Per protocol, eligible participants were randomized to one of the maintenance treatment arms. Not all participants from the induction period continued into the randomized maintenance phase.)
Treated | 0 | 337 | 332
Received Second Course of Pembrolizumab | 0 | 7 | 13
Completed | 0 | 0 | 0
Not Completed | 0 | 337 | 335
Not completed — Participant Ongoing in Study | 0 | 100 | 97
Not completed — Withdrawal by Subject | 0 | 9 | 3
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Death | 0 | 228 | 234

BASELINE CHARACTERISTICS:
Population: Pembrolizumab + Pemetrexed + Platinum Therapy (Induction Phase): All participants allocated to the pembrolizumab + Pemetrexed + Platinum Therapy arm in the Induction phase but not randomized into the maintenance phase; Pembrolizumab + Olaparib (Maintenance Phase): All participants randomized to the Pembrolizumab + Olaparib arm post Induction Phase; Pembrolizumab + Pemetrexed (Maintenance Phase): All participants randomized to the Pembrolizumab + Pemetrexed arm post Induction Phase.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab + Pemetrexed + Platinum Therapy (Induction Phase) | Pembrolizumab + Olaparib (Maintenance Phase) | Pembrolizumab + Pemetrexed (Maintenance Phase) | Total
Number analyzed (Participants) | 331 | 337 | 335 | 1003
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.3 (9.4) | 61.6 (8.6) | 61.8 (9.8) | 62.3 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109 | 110 | 109 | 328
  Male | 222 | 227 | 226 | 675
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 59 | 50 | 67 | 176
  Not Hispanic or Latino | 246 | 263 | 253 | 762
  Unknown or Not Reported | 26 | 24 | 15 | 65
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 4 | 1 | 10
  Asian | 56 | 91 | 72 | 219
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2 | 4
  Black or African American | 9 | 4 | 8 | 21
  White | 236 | 218 | 234 | 688
  More than one race | 11 | 7 | 9 | 27
  Unknown or Not Reported | 14 | 11 | 9 | 34
Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) at Baseline of Maintenance Phase [Count of Participants; unit: Participants] — Participants were assessed for ECOG PS; Grade 0: Fully active, able to carry on all pre-disease performance without restriction; Grade 1: Restricted in physically strenuous activity but ambulatory & able to carry out work of a light or sedentary nature; Grade 2: Ambulatory & capable of all selfcare but unable to carry out any work activities, up & about more than 50% of waking hours; Grade 3: Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours; Grade 4: Completely disabled, cannot carry on any selfcare, totally confined to bed or chair; Grade 5: Dead. Population: All participants randomized to the maintenance phase. Per protocol, data for this study specific baseline measure were not planned to be collected or reported for the induction phase.
  Participants
    number analyzed (Participants) | 0 | 337 | 335 | 672
    Grade 0 | 0 | 142 | 135 | 277
    Grade 1 | 0 | 195 | 200 | 395
Response at Baseline of Maintenance Phase [Count of Participants; unit: Participants] — Response per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) by blinded independent central review (BICR) consisted of Complete Response (CR)/Partial Response (PR) or Stable Disease (SD). CR: Disappearance of all target lesions; PR: ≥30% decrease in the sum of diameters (SOD) of target lesions; SD: Neither sufficient shrinkage for PR nor sufficient increase for progressive disease (PD: ≥20% increase in the SOD of target lesions. In addition to the relative increase of 20% the sum must also demonstrate an absolute increase of ≥5 mm; appearance ≥1 new lesions is also PD). Population: All participants randomized to the maintenance phase. Per protocol, data for this study specific baseline measure were not planned to be collected or reported for the induction phase.
  Participants
    number analyzed (Participants) | 0 | 337 | 335 | 672
    Complete Response (CR)/Partial Response (PR) | 0 | 189 | 192 | 381
    Stable Disease (SD) | 0 | 148 | 143 | 291
Programmed Cell Death Ligand 1 (PD-L1) Status at Baseline of Maintenance Phase [Count of Participants; unit: Participants] — Participants were assessed for their PD-L1 tumor expression level by immunohistochemistry assay using tumor tissue from a newly obtained biopsy. Participants with a tumor proportion score (TPS) ≥50% were classified as PD-L1 strongly positive and participants with a TPS <50% were classified as not strongly positive. Population: All participants randomized to the maintenance phase. Per protocol, data for this study specific baseline measure were not planned to be collected or reported for the induction phase.
  Participants
    number analyzed (Participants) | 0 | 337 | 335 | 672
    TPS<50% | 0 | 228 | 223 | 451
    TPS ≥50% | 0 | 109 | 110 | 219
    Not Evaluable | 0 | 0 | 1 | 1
    Missing | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time from randomization to the first documented progressive disease (PD) per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) based on blinded independent central review (BICR) or death due to any cause, whichever occurs first. PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD. PFS was analyzed by the non-parametric Kaplan-Meier (K-M) method. The protocol specified final analysis of PFS is presented here for the first pembrolizumab course in the Maintenance Phase. Per protocol, analysis for this outcome measure was not planned or conducted in the Induction Phase.
Time Frame: Up to ~31 months
Population: All randomized participants in the Maintenance Phase. Per protocol, analysis for this outcome measure was not planned or conducted in the Induction Phase.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Olaparib (Maintenance Phase) | Pembrolizumab + Pemetrexed (Maintenance Phase)
Number analyzed (Participants) | 337 | 335
Months | 7.1 [5.6 to 8.7] | 8.3 [6.9 to 11.5]
Statistical Analysis 1: Comparison: Pembrolizumab + Olaparib (Maintenance Phase) vs Pembrolizumab + Pemetrexed (Maintenance Phase); Test type: Superiority; p = 0.8721, Log Rank — One-sided p-value based on log-rank test stratified by Eastern Cooperative Oncology Group (ECOG) at pre-randomization visit, response at randomization and baseline PD-L1 status; Hazard Ratio (HR) = 1.12, 95% CI 2-sided [0.92 to 1.36] — Based on Cox regression model with Efron's method of tie handling and with treatment as a covariate stratified by ECOG at pre-randomization visit, response at randomization and baseline PD-L1 status

2. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to death due to any cause. OS was analyzed by the non-parametric K-M method. Participants without documented death at the time of analyses were censored at the date of last known to be alive. The protocol specified final analysis of OS is presented here for the first pembrolizumab course in the Maintenance Phase. Per protocol, analysis for this outcome measure was not planned or conducted in the Induction Phase.
Time Frame: Up to ~51 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Olaparib (Maintenance Phase) | Pembrolizumab + Pemetrexed (Maintenance Phase)
Number analyzed (Participants) | 337 | 335
Months | 20.7 [18.0 to 24.8] | 23.0 [19.0 to 26.4]
Statistical Analysis 1: Comparison: Pembrolizumab + Olaparib (Maintenance Phase) vs Pembrolizumab + Pemetrexed (Maintenance Phase); Test type: Superiority; p = 0.6649, Log Rank — One-sided p-value based on log-rank test stratified by ECOG at pre-randomization visit, response at randomization and baseline PD-L1 status; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.87 to 1.25] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Number of Participants Who Experience One or More Adverse Events (AEs)
Description: An AE is defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experience one or more AEs will be reported. The protocol specified final analysis will be presented for the first pembrolizumab course.
Time Frame: Up to ~5 years
Reporting Status: Not Posted, anticipated posting 2026-12

4. Secondary Outcome: Number of Participants Who Discontinue Study Treatment Due to an AE
Description: An AE is defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinue study treatment due to an AE will be reported. The protocol specified final analysis will be presented for the first pembrolizumab course.
Time Frame: Up to ~5 years
Reporting Status: Not Posted, anticipated posting 2026-12

5. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 (QLQ-C30) Global Health Status / Quality of Life (Items 29 and 30) Scale Score
Description: EORTC QLQ-C30 is a questionnaire to assess the overall quality of life (QoL) of cancer patients. Participant responses to questions regarding Global Health Status (GHS; "How would you rate your overall health during the past week?") and QoL ("How would you rate your overall quality of life during the past week?") are scored on a 7-point scale (1= Very poor to 7=Excellent). The combined score of GHS (Item 29) and QoL (Item 30) is computed by averaging the raw scores of the 2 items and then applying a linear transformation to standardize the average score, so that the combined scores range from 0-100. A higher score indicates a better outcome. The change from baseline in GHS and QoL combined score is presented. The protocol specified final analysis for the first pembrolizumab course in the Maintenance Phase is reported. Per protocol, analysis for this outcome measure was not planned or conducted in the Induction Phase.
Time Frame: Baseline and Week 24
Population: All randomized participants in the Maintenance Phase who received at least one dose of Maintenance Phase study treatment and had at least 1 patient reported outcome (PRO) assessment available. Per protocol, analysis for this outcome measure was not planned or conducted in the Induction Phase.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Pembrolizumab + Olaparib (Maintenance Phase) | Pembrolizumab + Pemetrexed (Maintenance Phase)
Number analyzed (Participants) | 337 | 332
Scores on a scale | -5.34 [-7.78 to -2.90] | -3.44 [-5.90 to -0.98]
Statistical Analysis 1: Comparison: Pembrolizumab + Olaparib (Maintenance Phase) vs Pembrolizumab + Pemetrexed (Maintenance Phase); Test type: Superiority; p = 0.2533, t-test, 2 sided — Two-sided p-value based on t test; Difference in Least Squares (LS) Means = -1.90, 95% CI 2-sided [-5.16 to 1.36] — Based on constrained longitudinal data analysis model (cLDA) model with PRO scores as response variable with covariates for treatment by time interaction, stratification factors, response at randomization and baseline PD-L1 expression as covariates

6. Secondary Outcome: Time to True Deterioration (TTD) in EORTC QLQ-C30 Global Health Status / Quality of Life (Items 29 & 30) Scale Score
Description: EORTC QLQ-C30 is a questionnaire to assess QoL of cancer patients. Participant responses to questions on GHS ("How would you rate your overall health during the past week?") and QoL ("How would you rate your overall QoL during the past week?") are scored on a 7-point scale (1= Very poor to 7=Excellent). The combined score of GHS (Item 29) and QoL (Item 30) is computed by averaging raw scores of the 2 items and applying a linear transformation to standardize the average score, so that the combined scores range from 0-100. A higher score indicates a better outcome. TTD is defined as the time from baseline to first onset of ≥10-point negative change (decrease) from baseline in GHS-QoL combined score. TTD estimated by non-parametric K-M method is presented here. A longer TTD indicates a better outcome. The protocol specified final analysis for the first pembrolizumab course in the Maintenance Phase is reported. Per protocol, analysis for this outcome was not done in the Induction Phase.
Time Frame: Up to ~24 months
Population: All randomized participants in the Maintenance Phase who received at least one dose of Maintenance Phase study treatment, had at least 1 PRO assessment and had data available for this EORTC QLQ-C30 outcome measure. Per protocol, analysis for this outcome was not planned or conducted in the Induction Phase.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Olaparib (Maintenance Phase) | Pembrolizumab + Pemetrexed (Maintenance Phase)
Number analyzed (Participants) | 329 | 316
Months | 19.81 [15.97 to NA] — Upper limit not reached at time of data cut-off due to insufficient number of participants with an event. | 17.28 [9.46 to NA] — Upper limit not reached at time of data cut-off due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Pembrolizumab + Olaparib (Maintenance Phase) vs Pembrolizumab + Pemetrexed (Maintenance Phase); Test type: Superiority; p = 0.8125, Log Rank — Two-sided p-value based on log-rank test stratified by ECOG at pre-randomization visit, response at randomization, and baseline PD-L1 expression; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.76 to 1.24] — Based on Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by ECOG at pre-randomization visit, response at randomization, and baseline PD-L1 expression

7. Secondary Outcome: Change From Baseline in EORTC Quality of Life Questionnaire Lung Cancer Module 13 (QLQ-LC13) Cough (Item 1) Scale Score
Description: EORTC QLQ-LC13 is a lung cancer specific questionnaire. Participant responses to the question regarding cough (Item 1): "How much did you cough?" are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0-100. A lower score indicates a better outcome. The change from baseline in EORTC QLQ-LC13 cough (Item 1) score is presented. The protocol specified final analysis for the first pembrolizumab course in the Maintenance Phase is reported. Per protocol, analysis for this outcome measure was not planned or conducted in the Induction Phase.
Time Frame: Baseline and Week 24
Population: All randomized participants in the Maintenance Phase who received at least one dose of Maintenance Phase study treatment and had at least 1 PRO assessment available. Per protocol, analysis for this outcome measure was not planned or conducted in the Induction Phase.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Pembrolizumab + Olaparib (Maintenance Phase) | Pembrolizumab + Pemetrexed (Maintenance Phase)
Number analyzed (Participants) | 337 | 332
Scores on a scale | -1.98 [-4.90 to 0.94] | -1.82 [-4.77 to 1.12]
Statistical Analysis 1: Comparison: Pembrolizumab + Olaparib (Maintenance Phase) vs Pembrolizumab + Pemetrexed (Maintenance Phase); Test type: Superiority; p = 0.9364, t-test, 2 sided — Two-sided p-value based on t test; Difference in LS Means = -0.16, 95% CI 2-sided [-4.02 to 3.71] — Based on cLDA model with the PRO scores as the response variable with covariates for treatment by time interaction, stratification factors, response at randomization, and baseline PD-L1 expression as covariates

8. Secondary Outcome: TTD in EORTC QLQ-LC13 Cough (Item 1) Scale Score
Description: EORTC QLQ-LC13 is a lung cancer specific questionnaire. Participant responses to the question regarding cough (Item 1): "How much did you cough?" are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0-100. A lower score indicates a better outcome. TTD is defined as the time from baseline to first onset of ≥10-point negative change (decrease) from baseline in cough (Item 1). TTD estimated by non-parametric K-M method is presented here. A longer TTD indicates a better outcome. The protocol specified final analysis for the first pembrolizumab course in the Maintenance Phase is reported. Per protocol, analysis for this outcome measure was not planned or conducted in the Induction Phase.
Time Frame: Up to ~24 months
Population: All randomized participants in the Maintenance Phase who received at least one dose of Maintenance Phase study treatment, had at least 1 PRO assessment and had data available for this EORTC QLQ-LC13 outcome measure. Per protocol, analysis for this outcome was not planned or conducted in the Induction Phase.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Olaparib (Maintenance Phase) | Pembrolizumab + Pemetrexed (Maintenance Phase)
Number analyzed (Participants) | 325 | 315
Months | NA [NA to NA] — Median, upper and lower limits not reached at time of data cut-off due to insufficient number of participants with an event. | NA [NA to NA] — Median, upper and lower limits not reached at time of data cut-off due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Pembrolizumab + Olaparib (Maintenance Phase) vs Pembrolizumab + Pemetrexed (Maintenance Phase); Test type: Superiority; p = 0.3782, Log Rank — [p-value comment as in outcome 6, analysis 1]; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.66 to 1.17] — [estimate comment as in outcome 6, analysis 1]

9. Secondary Outcome: Change From Baseline in EORTC QLQ-LC13 Chest Pain (Item 10) Scale Score
Description: EORTC QLQ-LC13 is a lung cancer specific questionnaire. Participant responses to the question regarding chest pain (Item 10): "Have you had pain in your chest?" are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A lower score indicates a better outcome. The change from baseline in EORTC QLQ-LC13 chest pain (Item 10) score is presented. The protocol specified final analysis for the first pembrolizumab course in the Maintenance Phase is reported. Per protocol, analysis for this outcome measure was not planned or conducted in the Induction Phase.
Time Frame: Baseline and Week 24
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Pembrolizumab + Olaparib (Maintenance Phase) | Pembrolizumab + Pemetrexed (Maintenance Phase)
Number analyzed (Participants) | 337 | 332
Scores on a scale | -0.82 [-3.25 to 1.61] | -0.47 [-2.92 to 1.98]
Statistical Analysis 1: Comparison: Pembrolizumab + Olaparib (Maintenance Phase) vs Pembrolizumab + Pemetrexed (Maintenance Phase); Test type: Superiority; p = 0.8285, t-test, 2 sided — Two-sided p-value based on t test; Difference in LS Means = -0.35, 95% CI 2-sided [-3.54 to 2.83] — [estimate comment as in outcome 7, analysis 1]

10. Secondary Outcome: TTD in EORTC QLQ-LC13 Chest Pain (Item 10) Scale Score
Description: EORTC QLQ-LC13 is a lung cancer specific questionnaire. Participant responses to the question regarding chest pain (Item 10): "Have you had pain in your chest?" are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A lower score indicates a better outcome. TTD is defined as the time from baseline to first onset of ≥10-point negative change (decrease) from baseline in chest pain (Item 10). TTD estimated by non-parametric K-M method is presented here. A longer TTD indicates a better outcome. The protocol specified final analysis for the first pembrolizumab course in Maintenance Phase is reported. Per protocol, analysis for this outcome measure was not planned or conducted in the Induction Phase.
Time Frame: Up to ~24 months
Population: All randomized participants in the Maintenance Phase who received at least one dose of Maintenance Phase study treatment, had at least 1 PRO assessment and had EORTC QLQ-LC13 data available for this outcome measure. Per protocol, analysis for this outcome was not planned or conducted in the Induction Phase.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Olaparib (Maintenance Phase) | Pembrolizumab + Pemetrexed (Maintenance Phase)
Number analyzed (Participants) | 325 | 315
Months | NA [NA to NA] — Median, upper and lower limits not reached at time of data cut-off due to insufficient number of participants with an event. | NA [NA to NA] — Median, upper and lower limits not reached at time of data cut-off due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Pembrolizumab + Olaparib (Maintenance Phase) vs Pembrolizumab + Pemetrexed (Maintenance Phase); Test type: Superiority; p = 0.6272, Log Rank — [p-value comment as in outcome 6, analysis 1]; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [0.78 to 1.51] — [estimate comment as in outcome 6, analysis 1]

11. Secondary Outcome: Change From Baseline in EORTC QLQ-C30 Dyspnea (Item 8) Scale Score
Description: EORTC QLQ-C30 is a questionnaire to assess the overall QoL of cancer patients. Participant responses to the question regarding dyspnea (Item 8): "Were you short of breath?" are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A lower score indicates a better outcome. The change from baseline in EORTC QLQ-C30 dyspnea (Item 8) score is presented. The protocol specified final analysis for the first pembrolizumab course in Maintenance Phase is reported. Per protocol, analysis for this outcome measure was not planned or conducted in the Induction Phase.
Time Frame: Baseline and Week 24
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Pembrolizumab + Olaparib (Maintenance Phase) | Pembrolizumab + Pemetrexed (Maintenance Phase)
Number analyzed (Participants) | 337 | 332
Scores on a scale | -0.16 [-3.07 to 2.76] | 1.35 [-1.60 to 4.31]
Statistical Analysis 1: Comparison: Pembrolizumab + Olaparib (Maintenance Phase) vs Pembrolizumab + Pemetrexed (Maintenance Phase); Test type: Superiority; p = 0.4422, t-test, 2 sided — Two-sided p-value based on t test; Difference in LS Means = -1.51, 95% CI 2-sided [-5.38 to 2.35] — [estimate comment as in outcome 7, analysis 1]

12. Secondary Outcome: TTD in EORTC QLQ-C30 Dyspnea (Item 8) Scale Score
Description: EORTC QLQ-C30 is a questionnaire to assess the overall QoL of cancer patients. Participant responses to the question regarding dyspnea (Item 8): "Were you short of breath?" are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A lower score indicates a better outcome. TTD is defined as the time from baseline to first onset of ≥10-point negative change (decrease) from baseline in dyspnea (Item 8). TTD estimated by non-parametric K-M method is presented here. A longer TTD indicates a better outcome. The protocol specified final analysis for the first pembrolizumab course in the Maintenance Phase is reported. Per protocol, analysis for this outcome measure was not planned or conducted in the Induction Phase.
Time Frame: Up to ~24 months
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Olaparib (Maintenance Phase) | Pembrolizumab + Pemetrexed (Maintenance Phase)
Number analyzed (Participants) | 329 | 316
Months | NA [NA to NA] — Median, upper and lower limits not reached at time of data cut-off due to insufficient number of participants with an event. | NA [NA to NA] — Median, upper and lower limits not reached at time of data cut-off due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Pembrolizumab + Olaparib (Maintenance Phase) vs Pembrolizumab + Pemetrexed (Maintenance Phase); Test type: Superiority; p = 0.9156, Log Rank — [p-value comment as in outcome 6, analysis 1]; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.74 to 1.31] — [estimate comment as in outcome 6, analysis 1]

13. Secondary Outcome: Change From Baseline in EORTC QLQ-C30 Physical Functioning (Items 1 to 5) Scale Score
Description: EORTC QLQ-C30 is a questionnaire to assess the overall QoL of cancer patients. Participant responses to 5 questions about their physical functioning (Items 1 to 5) are scored on a 4-point scale (1=Not at All to 4=Very Much). The combined score of items 1 to 5 is computed by averaging the raw scores of the 5 items and then applying a linear transformation to standardize the average score, so that the combined scores range from 0-100. A higher score indicates a better outcome. The change from baseline in EORTC QLQ-C30 physical functioning (Items 1-5) combined score is presented. The protocol specified final analysis for the first pembrolizumab course in Maintenance Phase is reported. Per protocol, analysis for this outcome measure was not planned or conducted in the Induction Phase.
Time Frame: Baseline and Week 24
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Pembrolizumab + Olaparib (Maintenance Phase) | Pembrolizumab + Pemetrexed (Maintenance Phase)
Number analyzed (Participants) | 337 | 332
Scores on a scale | -2.79 [-4.92 to -0.65] | -2.78 [-4.93 to -0.62]
Statistical Analysis 1: Comparison: Pembrolizumab + Olaparib (Maintenance Phase) vs Pembrolizumab + Pemetrexed (Maintenance Phase); Test type: Superiority; p = 0.9962, t-test, 2 sided — Two-sided p-value based on t test; Difference in LS Means = -0.01, 95% CI 2-sided [-2.94 to 2.93] — [estimate comment as in outcome 7, analysis 1]

14. Secondary Outcome: TTD in EORTC QLQ-C30 Physical Functioning (Items 1 to 5) Scale Score
Description: EORTC QLQ-C30 is a questionnaire to assess the overall QoL of cancer patients. Participant responses to 5 questions about their physical functioning (Items 1 to 5) are scored on a 4-point scale (1=Not at All to 4=Very Much). The combined score of items 1 to 5 is computed by averaging the raw scores of the 5 items and then applying a linear transformation to standardize the average score, so that the combined scores range from 0-100. A higher score indicates a better outcome. TTD is defined as the time from baseline to first onset of ≥10-point negative change (decrease) from baseline in physical functioning (Items 1 to 5). TTD estimated by non-parametric K-M method is presented here. A longer TTD indicates a better outcome. The protocol specified final analysis for the first pembrolizumab course in the Maintenance Phase is reported. Per protocol, analysis for this outcome measure was not planned or conducted in the Induction Phase.
Time Frame: Up to ~24 months
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Olaparib (Maintenance Phase) | Pembrolizumab + Pemetrexed (Maintenance Phase)
Number analyzed (Participants) | 329 | 316
Months | 20.96 [13.34 to NA] — Upper limit not reached at time of data cut-off due to insufficient number of participants with an event. | NA [17.28 to NA] — Median and upper limit not reached at time of data cut-off due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Pembrolizumab + Olaparib (Maintenance Phase) vs Pembrolizumab + Pemetrexed (Maintenance Phase); Test type: Superiority; p = 0.5517, Log Rank — [p-value comment as in outcome 6, analysis 1]; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [0.83 to 1.40] — [estimate comment as in outcome 6, analysis 1]

ADVERSE EVENTS:
Time Frame: Up to ~51 months
Description: All-cause Mortality (ACM): All enrolled participants; AEs: All participants who got ≥1 dose of study drug counted in the latest arm in which a participant got treated. Per protocol ACM and AEs were reported separately for pembrolizumab second course. Per protocol disease progression of cancer was not considered an AE unless related to study drug. Thus MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression", "Disease progression" unrelated to study drug are excluded as AEs
Groups:
- Pembrolizumab (First Course) + Olaparib (Maintenance Phase): Eligible participants with a complete/partial response or stable disease to treatment in the Induction Phase could enter Maintenance Phase. For the Maintenance Phase, participants received pembrolizumab 200 mg IV on Day 1 of each 3-week cycle for up to 31 cycles PLUS maintenance oral olaparib 300 mg twice daily. In the Maintenance Phase, participants continued to receive maintenance olaparib until progressive disease or toxicity. Across both phases, participants could receive pembrolizumab for a total treatment duration of up to ~35 cycles (up to ~2 years [cycle = 3 weeks]).
- Pembrolizumab (First Course) + Pemetrexed (Maintenance Phase): Eligible participants with a complete/partial response or stable disease to treatment in the Induction Phase could enter the Maintenance Phase. For the Maintenance Phase, participants received pembrolizumab 200 mg IV on Day 1 of each 3-week cycle for up to 31 cycles PLUS maintenance pemetrexed 500 mg/m^2 IV on Day 1 of each 3-week cycle. In the Maintenance Phase, participants continued to receive maintenance pemetrexed until progressive disease or toxicity. Across both phases, participants could receive pembrolizumab for a total treatment duration of up to ~35 cycles (up to ~2 years [cycle = 3 weeks]).
- Pembrolizumab (Second Course) + Olaparib (Maintenance Phase): In the Maintenance Phase, qualified participants who received pembrolizumab (200 mg IV on Day 1 of each 3-week cycle) plus olaparib (300 mg orally twice daily until progressive disease or toxicity) and who completed up to ~35 cycles of pembrolizumab (up to ~2 years [cycle =3 weeks]) may have been eligible to receive a second course of pembrolizumab at the same dose and schedule (200 mg on Day 1 of each 3-week cycle) for up to ~17 cycles (up to ~1 additional year).
- Pembrolizumab (Second Course) + Pemetrexed (Maintenance Phase): In the Maintenance Phase, qualified participants who received pembrolizumab (200 mg IV on Day 1 of each 3-week cycle) plus pemetrexed (500 mg/m^2 IV on Day 1 of each 3-week cycle until progressive disease or toxicity) and who completed up to ~35 cycles of pembrolizumab (up to ~2 years [cycle =3 weeks]) may have been eligible to receive a second course of pembrolizumab at the same dose and schedule (200 mg on Day 1 of each 3-week cycle) for up to ~17 cycles (up to ~1 additional year).
Arm/Group | Pembrolizumab + Pemetrexed + Platinum Therapy (Induction Phase) | Pembrolizumab (First Course) + Olaparib (Maintenance Phase) | Pembrolizumab (First Course) + Pemetrexed (Maintenance Phase) | Pembrolizumab (Second Course) + Olaparib (Maintenance Phase) | Pembrolizumab (Second Course) + Pemetrexed (Maintenance Phase)
All-Cause Mortality (participants affected / at risk) | 116/1003 | 233/337 | 233/335 | 0/7 | 2/13
Serious Adverse Events (participants affected / at risk) | 235/1003 | 118/337 | 125/332 | 0/7 | 1/13
Other Adverse Events (participants affected / at risk) | 872/1003 | 298/337 | 289/332 | 2/7 | 9/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + Pemetrexed + Platinum Therapy (Induction Phase) (N=1003) | Pembrolizumab (First Course) + Olaparib (Maintenance Phase) (N=337) | Pembrolizumab (First Course) + Pemetrexed (Maintenance Phase) (N=332) | Pembrolizumab (Second Course) + Olaparib (Maintenance Phase) (N=7) | Pembrolizumab (Second Course) + Pemetrexed (Maintenance Phase) (N=13)
Anaemia (Blood and lymphatic system disorders) | 24 (25) | 9 (9) | 8 (8) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 11 (11) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 7 (8) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 11 (14) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 18 (22) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 2 (2) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Hypophysitis (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Duodenal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal toxicity (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal wall thickening (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Jejunal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (6) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Noninfective sialoadenitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proctitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 8 (8) | 3 (3) | 5 (5) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 8 (8) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hyperthermia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 9 (9) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Serositis (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sudden death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Hepatitis toxic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated cholangitis (Hepatobiliary disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bacterial sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bronchopulmonary aspergillosis allergic (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 6 (6) | 2 (2) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 9 (9) | 6 (6) | 17 (18) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dengue fever (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Empyema (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Gangrene (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Giardiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pleural infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 23 (23) | 14 (16) | 11 (11) | 0 (0) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Pneumonia pseudomonal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 11 (11) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Serratia infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Severe acute respiratory syndrome (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suspected COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Testicular abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urethritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 5 (6) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Craniofacial fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incision site pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Creatinine renal clearance decreased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Influenza A virus test positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (4) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Fistula (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myeloproliferative neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Brain injury (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Brain oedema (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebellar ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral haematoma (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dural arteriovenous fistula (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated encephalitis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukoencephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Speech disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Superior sagittal sinus thrombosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 3 (3) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular dementia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device dislocation (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alcoholism (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 6 (6) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Diabetic nephropathy (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Renal tubular necrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gynaecomastia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (5) | 5 (6) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 11 (12) | 1 (1) | 5 (5) | 0 (0) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 7 (7) | 10 (10) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 7 (7) | 0 (0) | 0 (0) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Euthanasia (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angiodysplasia (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aortic aneurysm rupture (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aortitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arterial thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subclavian artery embolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Superficial vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular occlusion (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Venous thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + Pemetrexed + Platinum Therapy (Induction Phase) (N=1003) | Pembrolizumab (First Course) + Olaparib (Maintenance Phase) (N=337) | Pembrolizumab (First Course) + Pemetrexed (Maintenance Phase) (N=332) | Pembrolizumab (Second Course) + Olaparib (Maintenance Phase) (N=7) | Pembrolizumab (Second Course) + Pemetrexed (Maintenance Phase) (N=13)
Anaemia (Blood and lymphatic system disorders) | 385 (432) | 122 (176) | 125 (199) | 1 (1) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 141 (208) | 48 (83) | 19 (41) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 17 (22) | 19 (31) | 14 (24) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 235 (371) | 57 (105) | 32 (60) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 114 (156) | 57 (93) | 35 (60) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 27 (27) | 35 (41) | 19 (20) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 6 (7) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 169 (199) | 21 (24) | 39 (52) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 101 (121) | 39 (63) | 35 (57) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 310 (485) | 81 (106) | 63 (167) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 83 (110) | 28 (42) | 24 (35) | 0 (0) | 0 (0)
Asthenia (General disorders) | 107 (141) | 31 (42) | 38 (60) | 0 (0) | 1 (1)
Chest pain (General disorders) | 28 (28) | 22 (22) | 20 (24) | 0 (0) | 0 (0)
Early satiety (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 140 (161) | 58 (72) | 54 (73) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 4 (4) | 2 (3) | 5 (5) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 23 (23) | 11 (11) | 49 (66) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 54 (62) | 36 (43) | 27 (48) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 4 (5) | 1 (1) | 4 (4) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2) | 29 (34) | 28 (28) | 1 (1) | 1 (1)
Rhinitis (Infections and infestations) | 2 (2) | 2 (5) | 2 (2) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 110 (122) | 31 (42) | 52 (97) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 81 (91) | 28 (38) | 55 (86) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 33 (35) | 10 (12) | 14 (19) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 35 (37) | 46 (63) | 40 (67) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 17 (17) | 4 (6) | 10 (14) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 29 (30) | 31 (39) | 18 (20) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 155 (190) | 52 (77) | 52 (79) | 0 (0) | 1 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 32 (32) | 12 (17) | 25 (33) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 24 (28) | 15 (29) | 14 (30) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 12 (13) | 9 (9) | 12 (15) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 30 (33) | 11 (16) | 19 (24) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 21 (24) | 9 (14) | 10 (12) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 34 (34) | 47 (60) | 35 (43) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 28 (30) | 31 (32) | 26 (32) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 14 (15) | 15 (18) | 18 (22) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 18 (20) | 19 (22) | 20 (23) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 34 (36) | 31 (35) | 27 (30) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 26 (33) | 18 (20) | 8 (12) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 36 (41) | 29 (36) | 29 (34) | 1 (1) | 1 (1)
Paraesthesia (Nervous system disorders) | 9 (9) | 6 (8) | 12 (13) | 0 (0) | 1 (1)
Affect lability (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 36 (36) | 33 (41) | 38 (48) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 54 (55) | 26 (27) | 42 (48) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 12 (14) | 10 (15) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 52 (54) | 32 (38) | 29 (39) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 75 (76) | 31 (37) | 37 (43) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 24 (26) | 11 (14) | 17 (18) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-10-17): https://cdn.clinicaltrials.gov/large-docs/23/NCT03976323/Prot_SAP_000.pdf